CLINICAL TRIAL: NCT06099834
Title: Evaluation of Osseointegration Process of Implants With Different Length And Diameter By Different Methods
Brief Title: Evaluation of Osseointegration Process of Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, Associate Prof Dr, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 256
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Dental Implant Failed; Osseointegration Failure of Dental Implant
Keywords: osseointegration; dental implant; mobility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient selection (Other): Patient selection criteria were as follows: absence of any systemic disease; not being in American Society of Anesthesiologists (ASA) Class 3 or 4 according to the ASA Physical Status Classification System (Doyle, 2017); being older than 20 years of age; the existence of panoramic and dental volumetric tomography images of the area to be implanted; the presence of a suitable recipient bone for implantation with dental implants of the desired length and diameter.
  Interventions: Other: Patients selection
- Dental Implant Application (Other): Bredent SKY® dental implants were applied at a torque level of 30 N.cm as recommended by the manufacturer. The surgery and all measurements were performed by the same surgeon.
  Interventions: Other: Implnat placement
- Osseointegration and periodontal measurements (Other): Following the operations, the stability of the dental implants was measured at the 1st (T1), 4th (T4), and 12th (T12) weeks using Periotest (Periotest M, Modautal/Germany) and Osstell (Osstell AB-W&H, Sweden) devices. In accordance with the manufacturers' recommendations, the final implant stability quotient (ISQ) and Periotest values were determined by calculating the average of three measurements per implant. At the same time, periodontal index values of probing depth (PD-mm) and bleeding on probing (BOP-%) were recorded at the site of the dental implant at T4 and T12.
  Interventions: Other: Recall visits

INTERVENTIONS:
Other: Patients selection — Patient selection were selected according to selected criteria.
  Arms: Patient selection
Other: Implnat placement — dental implants were applied as recommended by the manufacturer.
  Arms: Dental Implant Application
Other: Recall visits — Following the operations, the stability of the dental implants was measured at the 1st (T1), 4th (T4), and 12th (T12) weeks using Periotest (Periotest M, Modautal/Germany) and Osstell (Osstell AB-W&H, Sweden) devices.
  Arms: Osseointegration and periodontal measurements

SUMMARY:
Implant stability is critical to successful osseointegration, the direct structural connection between the dental implant surface and bone. Implant stability must therefore be measured to evaluate implant success. The study evaluated the osseointegration of different sizes with two devices measuring stability with different methods.

DETAILED DESCRIPTION:
The 39 implants, 4.0 and 4.5 mm in diameter and 10 and 12 mm in length, in 19 patients were included. Hounsfield unit (HU) values obtained on cone beam computed tomography (CBCT) were recorded. Stabilities were measured with Periotest and resonance frequency analysis (RFA) at day 0 (intra-operative) and the 1st (T1), 4th (T4), and 12th (T12) weeks. Probing depth (PD) and bleeding on probing (BOP) scores were compared between T1 and T4.

ELIGIBILITY:
Inclusion Criteria:

* Absence of any systemic disease
* being older than 20 years of age
* having partial tooth deficiency in the posterior region of the lower jaw (molar tooth deficiency)
* having an indication for dental implant-supported fixed prosthesis
* at least 6 months had elapsed since the last tooth extraction in the area to be implanted
* having a soft tissue thickness of at least 1.5 mm and adherent gingival width of at least 2 mm
* the existence of panoramic and dental volumetric tomography images of the area to be implanted
* the presence of a suitable recipient bone for implantation with dental implants of the desired length and diameter
* completion of periodontal treatment and provision of oral hygiene training; and acceptable existing gingival health and oral hygiene for implant application (periodontally healthy) in the oral examinations performed following periodontal treatment.

Exclusion Criteria:

* being in American Society of Anesthesiologists (ASA) Class 3 or 4 according to the ASA Physical Status Classification System

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
RFA measurement | the 1st (T1), 4th (T4), and 12th (T12) weeks
  two SmartPeg transducers were used on each implant, and three measurements were completed: therefore, total number of registers was six for each implant. All assessment was carried out consecutively regardless register time or location. Measurements were completed by one only experienced dentist with knowl- edge of the Osstell ISQ system for RFA assessment
Periotest measurement | the 1st (T1), 4th (T4), and 12th (T12) weeks
  The periotest device is placed in a horizontal position 0.6-2 mm away from the tooth surface and two PTVs (PTV1 and PTV2) were calculated with a time difference of 20 min. During each measurement, the device delivers 16 impacts in 4 s to the object.

SECONDARY OUTCOMES:
Pocket probing depth | he 1st (T1), 4th (T4), and 12th (T12) weeks
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Abrahamsson I, Linder E, Lang NP. Implant stability in relation to osseointegration: an experimental study in the Labrador dog. Clin Oral Implants Res. 2009 Mar;20(3):313-8. doi: 10.1111/j.1600-0501.2008.01646.x. PMID 19405177
- [Background] Branemark PI, Hansson BO, Adell R, Breine U, Lindstrom J, Hallen O, Ohman A. Osseointegrated implants in the treatment of the edentulous jaw. Experience from a 10-year period. Scand J Plast Reconstr Surg Suppl. 1977;16:1-132. No abstract available. PMID 356184
- [Background] Boronat Lopez A, Balaguer Martinez J, Lamas Pelayo J, Carrillo Garcia C, Penarrocha Diago M. Resonance frequency analysis of dental implant stability during the healing period. Med Oral Patol Oral Cir Bucal. 2008 Apr 1;13(4):E244-7. PMID 18379449
- See also: for discussion — https://pubmed.ncbi.nlm.nih.gov/22669155/
- See also: for discussion — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4837777/